CLINICAL TRIAL: NCT06788093
Title: Reducing Overuse of Antibiotics With Decision Support in Lower Respiratory Tract Infections
Brief Title: Reducing Overuse of Antibiotics With Decision Support
Acronym: ROADS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Derek Williams, Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 240854; R01HS029331 (AHRQ)
Record Dates: First submitted 2024-07-16; First posted 2025-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lower Respiratory Tract Infection; Pneumonia; Asthma; Bronchiolitis, Viral
MeSH Terms: conditions — Pneumonia; Asthma; Bronchiolitis, Viral

STUDY DESIGN:
Intervention Model Description: In this pragmatic, randomized clinical trial, the investigators will evaluate the effectiveness and implementation of two stewardship-focused CDS interventions, alone and in combination, against usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care: Emergency Department (No Intervention): No experimental decision support will be provided to the emergency medicine providers in encounters randomized to the control arm. All patients will receive usual care and treatment will not be restricted or altered in any way by the study.
- CDS-ED (Experimental): The ED clinical decision support tool will be offered to emergency department providers in these enrolled encounters.
  Interventions: Behavioral: ED Clinical Decision Support (CDS-ED)
- Usual Care: Inpatient (No Intervention): No experimental decision support will be provided to the inpatient/ICU providers in encounters randomized to the control arm. All patients will receive usual care and treatment will not be restricted or altered in any way by the study.
- CDS-Tr (Experimental): The Transitions clinical decision support tool will be offered to inpatient/ICU providers in these enrolled encounters.
  Interventions: Behavioral: Transitions Clinical Decision Support (CDS-Tr)

INTERVENTIONS:
Behavioral: ED Clinical Decision Support (CDS-ED) — The ED-CDS intervention is designed as a discrete decision support aid to influence initial antibiotic decision-making in the ED. This intervention will feature a clinician-facing LRTI dashboard for end-users that assimilates relevant clinical data (e.g., vital signs, select diagnostic tests, links to reference information) and offers tailored suggestions for antibiotic initiation, related diagnostic testing, and in those receiving antibiotics, preferred options and alternatives for antibiotic choice, route, dose, and duration.
  Arms: CDS-ED
Behavioral: Transitions Clinical Decision Support (CDS-Tr) — The CDS-Tr intervention is designed as a longitudinal decision support aid to influence initial and ongoing (i.e., continuation, discontinuation, escalation, or de-escalation) antibiotic decision-making in the hospital setting. This intervention will also feature the LRTI dashboard along with additional tailored suggestions and recommendations for antibiotic decision-making upon hospital admission, and for those receiving antibiotics, at the time of discharge. Additionally, CDS-Tr will be active at the time of any service transition (i.e., hospital to intensive care or vice versa) and at pre-specified time points (e.g., approximately 48 hours and 120 hours following ED triage for encounters remaining in the hospital).
  Arms: CDS-Tr

SUMMARY:
Eliminating inappropriate antibiotic use in pediatric lower respiratory tract infections (LRTI) is the central focus of this research. LRTIs (pneumonia, bronchiolitis, and infection-related exacerbations of asthma) account for nearly one-third of all emergency department (ED) visits and 40% of all infection-related hospitalizations in US children. LRTIs also account for more antibiotic use in children's hospitals than any other condition, despite most LRTIs being viral in nature. Inappropriate antibiotics are associated with substantial adverse effects. Accordingly, national guidelines strongly discourage routine antibiotic use for bronchiolitis and acute asthma and argue for significantly reducing antibiotic exposure (initiation, spectrum, and duration) in pneumonia.

To address the problem of inappropriate antibiotic use, hospital-based antimicrobial stewardship programs (ASPs) are now common nationwide, and these programs have demonstrated effectiveness in some hospital settings. Unfortunately, traditional ASP approaches do not translate well to the fast-paced and unpredictable ED environment, and hospital-based ASP resources are finite and not always immediately available.

Clinical decision support (CDS) embedded within the electronic health record (EHR) is a strategy that could address the ED antibiotic stewardship gap. Informed by a deep understanding of the key facilitators and barriers to using CDS to support appropriate antibiotic use in ED and hospital settings, the investigators have developed two stewardship-focused CDS interventions for pediatric LRTI. The overarching goal of this research is to rigorously evaluate the implementation and effectiveness of these CDS tools, alone and in combination, against usual care only in a pragmatic randomized clinical trial at 3 U.S. children's hospitals.

DETAILED DESCRIPTION:
This is a usual care-controlled superiority clinical trial platform designed to evaluate the effects of hospital-based CDS in the ED (CDS-ED) and after transitioning to the hospital setting (CDS-TR) on antibiotic prescribing and related clinical outcomes for child and adolescent LRTI encounters at 3 U.S. children's hospitals. The investigators hypothesize that both interventions will be superior to usual care and, among patients presenting in the ED and subsequently admitted to the hospital, the combined interventions (CDS-ED + CDS-TR) will be most effective overall. Randomization will occur sequentially in two stages corresponding to the ED CDS and Transitions CDS populations. The first stage of randomization will allocate qualifying ED encounters 1:1 to CDS-ED vs. usual care alone in the ED. The second stage of randomization will allocate participants requiring hospitalization (those discharged from the hospital are not eligible) 1:1 to CDS-TR vs. usual care at the time of admission. To minimize bias, the trial will be embedded within clinical care with minimal exclusions and disruption to usual care activities. Investigators will be blinded to study arm assignment, though blinding of treating clinicians is not possible due to the nature of the study. The trial will also evaluate process and implementation outcomes throughout the study period within the platform population. A formal interim analysis is not planned.

ELIGIBILITY:
Inclusion Criteria:

1. ED encounter or admission to an inpatient hospital team.
2. EHR-based positive screen for suspected LRTI, defined as a qualifying chief complaint (e.g., cough, shortness of breath, etc.), plus triage documentation of abnormal respiratory effort and/or cough.

Exclusion Criteria: None

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2800 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness: 10-day Longitudinal Antimicrobial Spectrum Index | 10 days
  The Antibiotic Spectrum Index (ASI) is a numerical metric which quantifies the relative breadth of antimicrobial activity of a given antibiotic medication. Tracking the 10-day trajectory of ASI will capture changes in antibiotic use resulting from changes in antibiotic initiation, spectrum of antibiotic activity, and duration of antibiotic use.
Primary Safety: Proportion of Participants Experiencing Escalation in Treatment | 10 days
  Treatment escalation will capture the escalation to higher level of care and/or antibiotic treatment strategy

SECONDARY OUTCOMES:
Effectiveness: Proportion of Participants Experiencing Reduction of ASI Score | 10 days
  De-escalation of antibiotic exposure intensity (1+ level decrease in daily antibiotic exposure intensity) for a duration of at least 72 hours during the first 10 days of treatment
Effectiveness: Total Treatment Duration | 42 days
  Days until cessation of antibiotic exposure (i.e., daily periods with an ASI score greater than 0) for the index encounter, inclusive of antibiotics received in the ED and hospital, as well as any additional days of antibiotics prescribed at discharge up to 42 days after enrollment.
Effectiveness: ASI per Exposure Day | 10 days
  The numerator is the cumulative ASI during the first 10 days of treatment (T0-T240) and the denominator is the number of days of antibiotic exposure (i.e., daily periods with an ASI score greater than 0) during this same period.
Safety: Need for Intensive Care | 42 days
  Use of intensive care at any point during index encounter
Safety: Need for Invasive Mechanical Ventilation or Shock Requiring Vasoactive Medications | 42 days
  Need for intubation and/or need for vasoactive medications to manage uncompensated shock at any point during the index encounter (excludes intubation or vasoactive medications used for or during planned procedures or surgical intervention)
Safety: 3- and 14-day ED Reutilization | 14 days
  Any ED revisit occurring within 72 and 336 hours of index discharge that does not result in hospitalization
Safety: 3- and 14-day Hospital Reutilization | 14 days
  Any re-hospitalization occurring within 72 and 336 hours of index discharge
Death within 14 days of index discharge | 14 days
  Death by any cause occurring: 1) during the index encounter; 2) within 14 days of the index discharge, or 3) reutilization occurring within 14 days of the index discharge and that results in death at any time during that encounter

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Williams, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Benioff Children's Hospital - Oakland, Oakland, California
  - Benioff Children's Hospital - San Francisco, San Francisco, California
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No